CLINICAL TRIAL: NCT04549675
Title: Sun Safe Partners Online: Pilot Randomized Controlled Clinical Trial
Brief Title: Couple-focused Intervention for Sun Protection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Chief, Behavioral Sciences Professor, Dept of Medicine, Robert Wood Johnson Medical School, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro20150001694; 131503 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Skin Cancer Prevention
Keywords: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Sun Safe Partners Online Intervention (Experimental): Web-based intervention called Sun Safe Partners Online. Website developed by the study team. Participants received individual username and password to login.
  Interventions: Behavioral: Sun Safe Partners Online
- Generic Online Sun Safety Information intervention (Active Comparator): Publicly online available skin cancer and sun protection information emailed to participants in 4 seperate email links.
  Interventions: Behavioral: Generic Online Sun Safety Information intervention

INTERVENTIONS:
Behavioral: Sun Safe Partners Online — Sun Safe Partners Online has 4 individual-focused modules and 4 couple-focused modules focusing on skin cancer prevention education and sun protection.
  Arms: Arm 1 Sun Safe Partners Online Intervention
Behavioral: Generic Online Sun Safety Information intervention — 4 links to sent to participants from (1) The Skin Cancer Foundation's Skin Cancer Prevention guidelines, (2) the Centers for Disease Control and Prevention's information on risk factors for skin cancer, (3) the American Academy of Dermatology's information on how to select an appropriate sunscreen, and (4) The Skin Cancer Foundation's information on sun protective clothing. Participants were emailed a link to one of the resources each week for 4 weeks.
  Arms: Generic Online Sun Safety Information intervention

SUMMARY:
The goal of this pilot study is to develop and test a couple-based intervention to increase sun protection practices. First, the investigators will develop the intervention website, Sun Safe Partners online. Next, the investigators will gather feedback and preferences for content in a small sample of couples who do not regularly engage in sun protection practices. The investigators will also gather preliminary information regarding the impact of the couple-based intervention.

DETAILED DESCRIPTION:
Aim 1: To develop and evaluate the feasibility of a couple-based sun protection intervention.

Aim 2: To examine the impact of the couple-based sun protection intervention on sun protection practices, individual attitudes, relationship perspective on sun protection, and couples' discussion with each other and their supportive communications about sun protection.

Aim 3: To develop and refine a SunSafe Partners online intervention. This process includes refining existing intervention content drawn from the first phase of this pilot research as well as formative and usability studies to obtain user-generated feedback on additional content and the approach.

Aim 4: To gather pilot data on participation in and evaluations of the Sun Safe partner's intervention from Aim 3.

Arm 1: Web-based intervention called Sun Safe Partners Online

Arm 2: Generic Online Sun Safety Information intervention- 4 links emailed to participants

ELIGIBILITY:
Inclusion Criteria:

1. Both partners age 18-75 years or 19-75 in Nebraska and Alabama given the age of majority in those states;
2. Married or co-habiting with a significant other for at least one year;
3. Partner 1 willing to to provide contact information for their spouse;
4. Partner 1 and spouse respond with never, rarely, sometimes, or often to question " When outdoors in warm weather, how often do participants protect their skin (by staying in the shade or covering your body with protective clothes or 30+ SPF sunscreen)?" Those who respond with always to this question will be excluded.
5. Partner 1 and spouse have an email account and internet access.

Exclusion Criteria:

Partner 1 and spouse/partner have a personal history of skin cancer (non-melanoma or melanoma)

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Sun Protection Behaviors | Baseline to 1 month FU survey
  Impact of Sun Safe Partners Online vs Generic Online intervention on Sun protection behavior measures. The Sun Habits survey asked participants to rate their frequency of 5 sun protection behaviors (sunscreen, hat, shirt with sleeves, long pants, and sunglasses) on warm sunny days (1=never to 5=always).
Sun Exposure | Baseline to 1 month FU survey
  Sun Exposure: The Sun Habits Survey asked participants to rate the duration of outdoor time during peak hours on weekends and weekdays over the past summer months, 1=30 min or less, and 8=more than 6 hours. Self-report measures of time outdoors have s

OTHER OUTCOMES:
Perceived Risk of Skin cancer | Baseline to 1 month fu survey
  Three items assessed the perceived risk of skin cancer (sample item: "If I don't protect myself from the sun, I would feel vulnerable to getting skin cancer in my lifetime"). Items were rated on Likert-type response scales, ranging from 1 (strongly disagree) to 5 (strongly agree)
Sun Protection benefits | Baseline to 1 month fu survey
  Nine item scale assessessing sun protection benefits (sample item: "Regularly wearing sunscreen when in the sun would reduce my chances of getting skin cancer"). Scale utilizes likert items on 1 (strongly disagree) to 5 (strongly agree) scale.
Barriers to Sunscreen | Baseline to 1 month fu survey
  9 item scale measuring sunscreen barriers (sample item: "For me, using sunscreen when I am outside on a warm sunny day is not part of my daily routine"). Scale utilizes likert items on 1 (strongly disagree) to 5 (strongly agree) scale.
Barriers to sun protective clothing | Baseline to 1 month fu survey
  7 item scale measuring sunscreen barriers (sample item: ""For me, using sunscreen when I am outside on a warm sunny day is not part of my daily routine""). Scale utilizes likert items on 1 (strongly disagree) to 5 (strongly agree) scale.
Self-efficacy for sun protection | Baseline to 1 month FU survey
  9 item scale assessing confidence in performing sun protection behaviors. Sample item: "Are participants confident that they can use sunscreen on every part of their body that is not covered by clothing?" Scale utilizes likert items from 1 (not at all confident) to 5 (very confident).

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Manne S, Buller D, Devine K, Heckman C, Pagoto S, Frederick S, Mitarotondo A. Sun Safe Partners Online: Pilot Randomized Controlled Clinical Trial. J Med Internet Res. 2020 Sep 17;22(9):e18037. doi: 10.2196/18037. PMID 32673215